CLINICAL TRIAL: NCT01125059
Title: The Effect of Methadone on Perioperative Analgesia After Posterior Lumbar Fusion - A Randomized, Placebo-controlled, Double-blinded Study
Brief Title: Methadone Versus Placebo in Spine Fusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to fulfill recruitment
Sponsor: Northwestern University (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Dhanesh Gupta, Associate Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00027431
Record Dates: First submitted 2010-05-11; First posted 2010-05-18 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Pain
Keywords: hydromorphone; lumbar posterior spinal fusion; lumbosacral spondylosis; Spinal Fusion
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone Group (Active Comparator): 0.2 mg/kg IV methadone
  Interventions: Drug: Methadone
- Placebo Group (Placebo Comparator): 5 mL saline bolus
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Methadone — 0.2 mg/kg methadone IV bolus
  Other Names: Dolophine
  Arms: Methadone Group
Drug: Saline — 3 mL saline IV bolus
  Other Names: 0.9 NaCl
  Arms: Placebo Group

SUMMARY:
What is the influence of methadone on postoperative analgesia after lumbar interbody fusion in opioid naïve patients or patients who are taking less than equivalent of 15 mg IV morphine each day? What is the incidence of opioid related postoperative side effects after the administration of methadone in the operating room?

DETAILED DESCRIPTION:
Hypothesis:

1. We hypothesize that 0.2 mg/kg of methadone will result in decreased postoperative hydromorphone consumption compared to hydromorphone alone in opioid naïve patients or patients who are taking less than the equivalent of 15 mg IV morphine a day undergoing lumbar interbody fusion.
2. We hypothesize that the incidence of opioid related postoperative side effects will not be increased by the administration of methadone in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II, and III, male and non-pregnant female
* English-speaking patients
* Ages 18-75 years
* Undergoing elective one or two level posterior lumbar interbody fusion

Exclusion Criteria:

* Use of more than the equivalent of 15 mg of IV morphine/24 hr in the past 2 weeks.
* Use of drugs within the past 6 months that effect the pharmacokinetics or pharmacodynamics of opioids (i.e., benzodiazepines, anti-retroviral agents, rifampin, ketoconazole, erythromycin, or phenytoin).
* history of substance abuse at any time in the past
* known QT prolongation
* Non-elective operations (i.e., cancer or trauma)
* severe hepatic impairment (serum albumin < 3.0 g/dL in the presence of a history of liver disease)
* pregnancy
* inability to operate a patient-controlled analgesia device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Hydromorphone postoperative opioid consumption (POC) at 48 hours | 48 hrs
  PCA opioid consumption during the initial postoperative 48 hours after arriving in the PACU

SECONDARY OUTCOMES:
Intraoperative remifentanil consumption | the 8 hours prior to arrival in the recovery room
  intraoperative consumption of remifentanil--the amount of remifentanil used in the OR (i.e., the 2-8 hours prior to arrival in the recovery room)
pain at rest and with movement (numerical Rating Scale, NRS) | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs
the level of sedation (modified Observer's Assessment of Alertness and Sedation Scale, modified OAA/S scale) | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs
the number of occurrences of ventilatory depression during each evaluation interval | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs
number of occurrences of nausea (resulting in treatment) | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs
recorded emesis | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs
occurrence of pruritus | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs
Hydromorphone postoperative opioid consumption (POC) | 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs
  PCA opioid consumption at postoperative 1 hr, 6 hrs, 12 hrs, 24 hrs, 36 hrs after arriving in the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Dhanesh K Gupta, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Jadad AR, Browman GP. The WHO analgesic ladder for cancer pain management. Stepping up the quality of its evaluation. JAMA. 1995 Dec 20;274(23):1870-3. PMID 7500538
- [Background] Upton RN, Semple TJ, Macintyre PE. Pharmacokinetic optimisation of opioid treatment in acute pain therapy. Clin Pharmacokinet. 1997 Sep;33(3):225-44. doi: 10.2165/00003088-199733030-00005. PMID 9314613
- [Background] Taylor S, Kirton OC, Staff I, Kozol RA. Postoperative day one: a high risk period for respiratory events. Am J Surg. 2005 Nov;190(5):752-6. doi: 10.1016/j.amjsurg.2005.07.015. PMID 16226953
- [Background] Taylor S, Voytovich AE, Kozol RA. Has the pendulum swung too far in postoperative pain control? Am J Surg. 2003 Nov;186(5):472-5. doi: 10.1016/j.amjsurg.2003.07.021. PMID 14599609
- [Background] Liu N, Kuhlman G, Dalibon N, Moutafis M, Levron JC, Fischler M. A randomized, double-blinded comparison of intrathecal morphine, sufentanil and their combination versus IV morphine patient-controlled analgesia for postthoracotomy pain. Anesth Analg. 2001 Jan;92(1):31-6. doi: 10.1097/00000539-200101000-00007. PMID 11133596
- [Background] Joris J, Kaba A, Lamy M. Transition between anesthesia and post-operative analgesia: relevance of intra-operative administration of analgesics. Acta Anaesthesiol Belg. 2001;52(3):271-9. PMID 11732383
- [Background] Carroll IR, Angst MS, Clark JD. Management of perioperative pain in patients chronically consuming opioids. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):576-91. doi: 10.1016/j.rapm.2004.06.009. PMID 15635517
- [Background] Yaksh TL, Hua XY, Kalcheva I, Nozaki-Taguchi N, Marsala M. The spinal biology in humans and animals of pain states generated by persistent small afferent input. Proc Natl Acad Sci U S A. 1999 Jul 6;96(14):7680-6. doi: 10.1073/pnas.96.14.7680. PMID 10393880
- [Background] Parker RK, Holtmann B, White PF. Effects of a nighttime opioid infusion with PCA therapy on patient comfort and analgesic requirements after abdominal hysterectomy. Anesthesiology. 1992 Mar;76(3):362-7. doi: 10.1097/00000542-199203000-00007. PMID 1539846
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Chui PT, Gin T. A double-blind randomised trial comparing postoperative analgesia after perioperative loading doses of methadone or morphine. Anaesth Intensive Care. 1992 Feb;20(1):46-51. doi: 10.1177/0310057X9202000109. PMID 1609941
- [Background] Egan TD, Huizinga B, Gupta SK, Jaarsma RL, Sperry RJ, Yee JB, Muir KT. Remifentanil pharmacokinetics in obese versus lean patients. Anesthesiology. 1998 Sep;89(3):562-73. doi: 10.1097/00000542-199809000-00004. PMID 9743391
- [Background] Lemmens HJ, Brodsky JB, Bernstein DP. Estimating ideal body weight--a new formula. Obes Surg. 2005 Aug;15(7):1082-3. doi: 10.1381/0960892054621350. PMID 16105412
- [Background] Bowdle TA, Even A, Shen DD, Swardstrom M. Methadone for the induction of anesthesia: plasma histamine concentration, arterial blood pressure, and heart rate. Anesth Analg. 2004 Jun;98(6):1692-1697. doi: 10.1213/01.ANE.0000114085.20751.20. PMID 15155330
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Apfelbaum JL, Gan TJ, Zhao S, Hanna DB, Chen C. Reliability and validity of the perioperative opioid-related symptom distress scale. Anesth Analg. 2004 Sep;99(3):699-709. doi: 10.1213/01.ANE.0000133143.60584.38. PMID 15333398
- [Background] van Dorp EL, Kest B, Kowalczyk WJ, Morariu AM, Waxman AR, Arout CA, Dahan A, Sarton EY. Morphine-6beta-glucuronide rapidly increases pain sensitivity independently of opioid receptor activity in mice and humans. Anesthesiology. 2009 Jun;110(6):1356-63. doi: 10.1097/ALN.0b013e3181a105de. PMID 19461298